CLINICAL TRIAL: NCT00790296
Title: A Pilot, Randomized Double-Blind Placebo-Controlled Crossover Study of Synthetic Thyrotropin Releasing Hormone (TRH) Administration for the Treatment of Fatigue in Patients With Cancer
Brief Title: Evaluation of Synthetic Thyrotropin Releasing Hormone (TRH) as a Treatment for Cancer-related Fatigue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analyses showed statistically and clinically significant results.
Sponsor: UConn Health (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Hollfelder foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 05-269-2; 601
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cancer-related Fatigue
Keywords: cancer fatigue
MeSH Terms: interventions — Thyrotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thyrotropin releasing hormone (TRH) (Experimental): TRH
  Interventions: Drug: Thyrotropin releasing hormone (TRH)
- Saline (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thyrotropin releasing hormone (TRH) — 0.5mg and 1.5mg
  Arms: Thyrotropin releasing hormone (TRH)
Drug: Placebo — Saline
  Arms: Saline

SUMMARY:
The primary objective of the study is to evaluate thyrotropin releasing hormone (TRH) as a treatment for cancer-related fatigue.

The central hypothesis of this pilot study is that TRH is more efficacious than placebo in alleviating cancer-related fatigue in patients with breast or prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cancer who have undergone or are currently undergoing radiation or chemotherapy therapy and are expected not to have any significant change in cancer treatment sessions during the study period
* Provide written informed consent prior to initiation of any study-related procedures.
* Male or female, 18 years of age or older with a diagnosis of cancer.
* Able to understand and comply with the requirements of the study.

Exclusion criteria:

* Hospitalized patients.
* Patients with an identifiable diagnosis of substance abuse or dependence within 6 months prior to evaluation (except those in full remission, or those with caffeine or nicotine dependence) as defined by DSM-IV criteria.
* Patients with any of the following cardiovascular symptomatology.
* Office systolic BP > 160mmHg and/or diastolic BP > 90mmHg.
* Persons with a resting hear rate of > 100 beats per minute
* Persons with a history of chronic stable angina
* Persons with myocardial infarction or unstable angina or vascular surgery within 6 months
* Persons with history of vaso-vagal or other syncopal episodes
* Patients with any known clinically significant cardiac problems
* Patients with any history of stroke or at significant risk for stroke.
* Patients with a history of seizures
* Patients with a history of asthma
* Patients with any clinically significant unstable or inadequately treated co- morbid medical condition or patients currently on medications that would confound evaluation of CF (e.g. diabetes, CHF, history of other cancers) as judged by the investigator.
* Patients with any clinically significant, unstable psychiatric disorder (except mild to moderate depressive or anxiety disorders) or patients on psychotropic medications that would confound CF assessment as judged by the investigator. Patients with history of depressive or anxiety disorders will not be excluded from the study
* Patients with a history of illnesses or treatments that would be expected to significantly alter immune function (viz. HIV infection, systemic lupus erythematosus, patients taking immunosuppressive medications).
* Patients with diseases or on medications that significantly affect the hypothalamic-pituitary-adrenocortical (HPA) axis function (viz. Cushings disease).
* Pregnant patients, breastfeeding or plans to become pregnant during the study
* Patients with known allergy to TRH
* Any other condition, which, in the opinion of the investigator, would make the patient, unsuited for enrollment, confound CF evaluation or could interfere with the patient's participation in the study.
* Patients with medically reversible causes of CF (viz., anemia, hypothyroidism, electrolyte abnormalities etc).
* Patients with potentially treatable associated symptoms dominating the CF scenario such as pain, or sleep disturbances which may have a significant causal relationship to CF.
* Patients identified as pregnant based on the pregnancy test during screening.
* Patients physically unable to complete the walking test (WT) assessment or when the WT would increase risk for medical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Winokur, MD PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited per referrals from oncology clinics at UCHC and Gray Cancer Center at Hartford Hospital
Pre-assignment Details: Two participants signed informed consent but was not randomized as she did not meet study eligibility criteria
Groups:
- TRH Then Saline: TRH (0.5mg) given first followed by Saline
- Saline Then TRH: Saline given first followed by TRH (0.5 mg)
Period: Overall Study
Arm/Group | TRH Then Saline | Saline Then TRH
Started | 5 | 6
Completed | 4 | 4
Not Completed | 1 | 2
Not completed — Did not meet study eligibility criteria | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRH Then Saline | Saline Then TRH | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.4) | 58 (9.4) | 58 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale for Energy (VAS-E)Score From Baseline to 7 Hrs Post Study Medication Infusion
Description: 1 to 100 scale with 1 referring to No Energy and 100 referring to Normal Energy.
Time Frame: Baseline and 7 hours post study medication infusion
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Thyrotropin-releasing Hormone (TRH): TRH given as 0.5mg and 1.5mg intravenously
- Saline: Saline given Intravenously
Arm/Group | Thyrotropin-releasing Hormone (TRH) | Saline
Number analyzed (Participants) | 4 | 4
Scores on a scale | 14.67 (21.1) | -1.67 (16)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Thyrotropin-releasing Hormone (TRH) | Saline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Limitation: small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes